CLINICAL TRIAL: NCT03412071
Title: Testing the Ability of a Microbiome - Focused Intervention to Reduce HIV Susceptibility in Ugandan Men
Brief Title: Effect of Antibiotics on Penile Microbiome and HIV Susceptibility Study in Ugandan Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: UVRI-IAVI HIV Vaccine Program (Unknown); Entebbe General Hospital (Unknown)
Responsible Party: Principal Investigator, Rupert Kaul, Professor - Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Penile microbiome antibiotics
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Foreskin HIV Susceptibility
MeSH Terms: interventions — Tinidazole; Metronidazole; Clindamycin; Hydrogen Peroxide

STUDY DESIGN:
Intervention Model Description: Randomized, open label with 5 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (No Intervention): 25 HIV-uninfected, uncircumcised men will be immediately circumcised following enrollment. This group will serve as the comparison to the four intervention groups.
- Oral tinidazole group (Active Comparator): 25 HIV-uninfected, uncircumcised men will be randomized to receive oral tinidazole 2g once a day for two days.
  Interventions: Drug: Oral Tinidazole
- Topical metronidazole (0.75%) group (Active Comparator): 25 HIV-uninfected, uncircumcised men will be randomized to apply topical 0.75% metronidazole cream to the foreskin twice a day for one week, and then twice a week for three weeks.
  Interventions: Drug: Topical metronidazole
- Topical clindamycin (2%) group (Active Comparator): 25 HIV-uninfected, uncircumcised men will be randomized to apply topical 2% clindamycin cream to the foreskin twice a day for one week, and then twice a week for three weeks.
  Interventions: Drug: Topical Clindamycin
- Topical hydrogen peroxide (1%) group (Active Comparator): 25 HIV-uninfected, uncircumcised men will be randomized to apply 1% hydrogen peroxide cream to the foreskin twice a day for one week, and then twice a week for three weeks.
  Interventions: Drug: Topical Hydrogen Peroxide

INTERVENTIONS:
Drug: Oral Tinidazole — Please see description under arms
  Other Names: FASIGYN 500mgs
  Arms: Oral tinidazole group
Drug: Topical metronidazole — Please see description under arms
  Other Names: Rozex 0.75%
  Arms: Topical metronidazole (0.75%) group
Drug: Topical Clindamycin — Please see description under arms
  Other Names: Dalacin cream 2%
  Arms: Topical clindamycin (2%) group
Drug: Topical Hydrogen Peroxide — Please see description under arms
  Other Names: Crystacide 1%
  Arms: Topical hydrogen peroxide (1%) group

SUMMARY:
This pilot study will assess the impact of four antimicrobial products (3 topical, one systemic) on the foreskin microbiome and HIV susceptibility of foreskin-derived CD4+ T cells. Participants will include HIV-uninfected Ugandan men presenting for elective male circumcision to reduce their HIV risk.

DETAILED DESCRIPTION:
RATIONALE: The foreskin is the site of most HIV acquisition in uncircumcised heterosexual men, and male circumcision (MC) reduces HIV risk by almost 60%. However, cultural and practical barriers have led to suboptimal uptake. Foreskin inflammation, defined by elevated levels of pro-inflammatory cytokines in the prepuce, is a key determinant of HIV acquisition risk in uncircumcised men, and anaerobic bacteria within the foreskin microbiome may be an important cause of this inflammation.

OBJECTIVES: A pilot in vivo - in vitro clinical study of four potential interventions to reduce HIV susceptibility in the foreskin by altering the microbiome. The study is a collaboration between the University of Toronto, IAVI-UVRI, and the Entebbe General Hospital. We will recruit 125 men presenting for elective MC, along with regular female sexual partners (if applicable). Participants will be randomized (n=25 per group) to immediate MC, or to one of four intervention arms: twice-daily application of topical metronidazole 0.75%; twice-daily application of topical clindamycin 2%; twice daily application of hydrogen peroxide 1%; or oral tinidazole 2g once a day for two days. Swabs for immune and microbiome studies will be collected before and after product. After 4 weeks the MC procedure will be performed; foreskin CD4+ T cell susceptibility to HIV will be quantified using a flow cytometry-based pseudovirus assay, and tissue immunohistochemistry performed. The primary and secondary endpoints are outlined below. A secondary study will assess the impact of penile topical antibiotic application on immunology and the microbiome in the genital tract of female sexual partners.

OUTCOMES: This in vivo - in vitro clinical trial will define the causal role of the penile microbiome in HIV susceptibility, and will assess potential strategies to take forward into HIV efficacy trials in uncircumcised heterosexual men.

ELIGIBILITY:
Enrollment criteria include:

1. Aged 18 years or older
2. Biological male
3. Uncircumcised
4. HIV seronegative
5. Willing to comply with the requirements of the protocol
6. No current sexually transmitted infection (N. gonorrhoeae or C. trachomatis)
7. No clinically relevant genital symptoms / signs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Foreskin HIV susceptibility can only be assessed in biological males.
Enrollment: 125 (Estimated)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-12-07 (Estimated); Study Completion 2019-12-07 (Estimated)

PRIMARY OUTCOMES:
% HIV entry into foreskin derived CD4+ T cells | 4 weeks
  This measure will utilize a validated pseudovirus entry assay.

SECONDARY OUTCOMES:
Tissue density of HIV-susceptible CD4+ T cells | 4 weeks
  The density of CD4+ T cells in foreskin tissues will be assayed using immunohistochemistry, and the % pseudovirus entry (see primary endpoint, above) will be used to calculate the tissue density of HIV-susceptible CD4+ T cells.
CD4+ T cell subsets in foreskin tissue | 4 weeks
  Immunofluorescence microscopy (IF) will be used to quantify CD4+ T cell subsets foreskin tissue after circumcision.
Density of Langerhans cells in foreskin tissue | 4 weeks
  Immunofluorescence microscopy (IF) will be used to quantify Langerhans cells in foreskin tissue after circumcision.
Presence of foreskin inflammation | 4 weeks
  Cytokine/chemokines will be assayed by ELISA, and foreskin inflammation defined as the presence of ≥3/7 inflammatory cytokines within the top quartile for that cytokine.
Foreskin microbiome composition | 4 weeks
  The foreskin (prepuce) microbiome will be characterized based on 16S rRNA sequencing.
Foreskin tissue explant HIV susceptibility | 4 weeks
  Foreskin tissue susecptibility to HIV infection will be quantified, based on p24 ELISA after ex vivo incubation with a primary HIV isolate.

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Kaul, MD/PhD, Principal Investigator — University of Toronto; Ronald M Galiwango, MBChB/MSc, Study Director — University of Toronto
Locations (1):
- UVRI-IAVI HIV Vaccine Program, Entebbe, Wakiso, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gray RH, Wawer MJ, Kigozi G. Programme science research on medical male circumcision scale-up in sub-Saharan Africa. Sex Transm Infect. 2013 Aug;89(5):345-9. doi: 10.1136/sextrans-2012-050595. Epub 2013 May 22. PMID 23698513
- [Background] Liu CM, Hungate BA, Tobian AA, Serwadda D, Ravel J, Lester R, Kigozi G, Aziz M, Galiwango RM, Nalugoda F, Contente-Cuomo TL, Wawer MJ, Keim P, Gray RH, Price LB. Male circumcision significantly reduces prevalence and load of genital anaerobic bacteria. mBio. 2013 Apr 16;4(2):e00076. doi: 10.1128/mBio.00076-13. PMID 23592260
- [Background] Prodger JL, Gray R, Kigozi G, Nalugoda F, Galiwango R, Hirbod T, Wawer M, Hofer SO, Sewankambo N, Serwadda D, Kaul R. Foreskin T-cell subsets differ substantially from blood with respect to HIV co-receptor expression, inflammatory profile, and memory status. Mucosal Immunol. 2012 Mar;5(2):121-8. doi: 10.1038/mi.2011.56. Epub 2011 Nov 16. PMID 22089029
- [Background] Prodger JL, Gray RH, Shannon B, Shahabi K, Kong X, Grabowski K, Kigozi G, Nalugoda F, Serwadda D, Wawer MJ, Reynolds SJ, Liu CM, Tobian AA, Kaul R. Chemokine Levels in the Penile Coronal Sulcus Correlate with HIV-1 Acquisition and Are Reduced by Male Circumcision in Rakai, Uganda. PLoS Pathog. 2016 Nov 29;12(11):e1006025. doi: 10.1371/journal.ppat.1006025. eCollection 2016 Nov. PMID 27898732
- [Background] Prodger JL, Hirbod T, Kigozi G, Nalugoda F, Reynolds SJ, Galiwango R, Shahabi K, Serwadda D, Wawer MJ, Gray RH, Kaul R; Rakai Genital Immunology Research Group. Immune correlates of HIV exposure without infection in foreskins of men from Rakai, Uganda. Mucosal Immunol. 2014 May;7(3):634-44. doi: 10.1038/mi.2013.83. Epub 2013 Oct 23. PMID 24150258
- [Background] Menard JP. Antibacterial treatment of bacterial vaginosis: current and emerging therapies. Int J Womens Health. 2011;3:295-305. doi: 10.2147/IJWH.S23814. Epub 2011 Aug 23. PMID 21976983
- [Background] Rashed HT. Evaluation of the effect of hydrogen peroxide as a mouthwash in comparison with chlorhexidine in chronic periodontitis patients: A clinical study. J Int Soc Prev Community Dent. 2016 May-Jun;6(3):206-12. doi: 10.4103/2231-0762.183114. Epub 2016 May 30. PMID 27382535
- [Background] Armstrong NR, Wilson JD. Tinidazole in the treatment of bacterial vaginosis. Int J Womens Health. 2010 Aug 9;1:59-65. doi: 10.2147/ijwh.s4455. PMID 21072275
- [Background] Baggaley R, Doherty M, Ball A, Ford N, Hirnschall G. The Strategic Use of Antiretrovirals to Prevent HIV Infection: A Converging Agenda. Clin Infect Dis. 2015 Jun 1;60 Suppl 3:S159-60. doi: 10.1093/cid/civ091. PMID 25972496
- [Background] TenoRes Study Group. Global epidemiology of drug resistance after failure of WHO recommended first-line regimens for adult HIV-1 infection: a multicentre retrospective cohort study. Lancet Infect Dis. 2016 May;16(5):565-575. doi: 10.1016/S1473-3099(15)00536-8. Epub 2016 Jan 29. Erratum In: Lancet Infect Dis. 2016 Jun;16(6):636. doi: 10.1016/S1473-3099(16)30089-5. Lancet Infect Dis. 2018 Jan;18(1):21. doi: 10.1016/S1473-3099(17)30723-5. PMID 26831472
- [Background] Auvert B, Taljaard D, Lagarde E, Sobngwi-Tambekou J, Sitta R, Puren A. Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial. PLoS Med. 2005 Nov;2(11):e298. doi: 10.1371/journal.pmed.0020298. Epub 2005 Oct 25. PMID 16231970
- [Background] Bailey RC, Moses S, Parker CB, Agot K, Maclean I, Krieger JN, Williams CF, Campbell RT, Ndinya-Achola JO. Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial. Lancet. 2007 Feb 24;369(9562):643-56. doi: 10.1016/S0140-6736(07)60312-2. PMID 17321310
- [Background] Gray RH, Kigozi G, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chaudhary MA, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Williams CF, Opendi P, Reynolds SJ, Laeyendecker O, Quinn TC, Wawer MJ. Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial. Lancet. 2007 Feb 24;369(9562):657-66. doi: 10.1016/S0140-6736(07)60313-4. PMID 17321311
- [Background] Sgaier SK, Reed JB, Thomas A, Njeuhmeli E. Achieving the HIV prevention impact of voluntary medical male circumcision: lessons and challenges for managing programs. PLoS Med. 2014 May 6;11(5):e1001641. doi: 10.1371/journal.pmed.1001641. eCollection 2014 May. PMID 24800840
- [Background] Kigozi G, Wawer M, Ssettuba A, Kagaayi J, Nalugoda F, Watya S, Mangen FW, Kiwanuka N, Bacon MC, Lutalo T, Serwadda D, Gray RH. Foreskin surface area and HIV acquisition in Rakai, Uganda (size matters). AIDS. 2009 Oct 23;23(16):2209-13. doi: 10.1097/QAD.0b013e328330eda8. PMID 19770623
- [Background] Anahtar MN, Byrne EH, Doherty KE, Bowman BA, Yamamoto HS, Soumillon M, Padavattan N, Ismail N, Moodley A, Sabatini ME, Ghebremichael MS, Nusbaum C, Huttenhower C, Virgin HW, Ndung'u T, Dong KL, Walker BD, Fichorova RN, Kwon DS. Cervicovaginal bacteria are a major modulator of host inflammatory responses in the female genital tract. Immunity. 2015 May 19;42(5):965-76. doi: 10.1016/j.immuni.2015.04.019. PMID 25992865
- [Background] Bolduc JF, Ouellet M, Hany L, Tremblay MJ. Toll-Like Receptor 2 Ligation Enhances HIV-1 Replication in Activated CCR6+ CD4+ T Cells by Increasing Virus Entry and Establishing a More Permissive Environment to Infection. J Virol. 2017 Jan 31;91(4):e01402-16. doi: 10.1128/JVI.01402-16. Print 2017 Feb 15. PMID 27928019
- [Background] Esra RT, Olivier AJ, Passmore JA, Jaspan HB, Harryparsad R, Gray CM. Does HIV Exploit the Inflammatory Milieu of the Male Genital Tract for Successful Infection? Front Immunol. 2016 Jun 24;7:245. doi: 10.3389/fimmu.2016.00245. eCollection 2016. PMID 27446076
- [Background] Bukusi E, Thomas KK, Nguti R, Cohen CR, Weiss N, Coombs RW, Holmes KK. Topical penile microbicide use by men to prevent recurrent bacterial vaginosis in sex partners: a randomized clinical trial. Sex Transm Dis. 2011 Jun;38(6):483-9. PMID 22256334
- [Background] Jhingta P, Bhardwaj A, Sharma D, Kumar N, Bhardwaj VK, Vaid S. Effect of hydrogen peroxide mouthwash as an adjunct to chlorhexidine on stains and plaque. J Indian Soc Periodontol. 2013 Jul;17(4):449-53. doi: 10.4103/0972-124X.118315. PMID 24174723
- [Background] V Sgibnev A, A Kremleva E. Vaginal Protection by H2O2-Producing Lactobacilli. Jundishapur J Microbiol. 2015 Oct 17;8(10):e22913. doi: 10.5812/jjm.22913. eCollection 2015 Oct. PMID 26587206
- [Derived] Galiwango RM, Bagaya B, Mpendo J, Joag V, Okech B, Nanvubya A, Ssetaala A, Muwanga M, Kaul R. Protocol for a randomized clinical trial exploring the effect of antimicrobial agents on the penile microbiota, immunology and HIV susceptibility of Ugandan men. Trials. 2019 Jul 19;20(1):443. doi: 10.1186/s13063-019-3545-7. PMID 31324206